CLINICAL TRIAL: NCT00055133
Title: A Phase 2 Open-Label Clinical Study Using Intravenous Paxceed™ to Treat Patients With Rheumatoid Arthritis
Brief Title: A Study Using Intravenous Paxceed™ to Treat Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Angiotech Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 008-MPRA02
Record Dates: First submitted 2003-02-19; First posted 2003-02-21 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; Paxceed; Micellar Paclitaxel
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Injections

INTERVENTIONS:
Drug: Micellar Paclitaxel for Injection

SUMMARY:
Paxceed™ is being developed by Angiotech Pharmaceuticals, Inc. for the treatment of Rheumatoid Arthritis (RA). The main objective of this study is to determine the effectiveness of treatment with Paxceed™ in patients with RA. In RA, there is an increase in cell growth and changes in cell function. The active substance in Paxceed™, paclitaxel, has undergone clinical studies as a cancer chemotherapeutic agent and has demonstrated its usefulness as an agent that stops growth of cells and blocks certain types of cell function associated with RA. Because of these effects, it is thought that Paxceed™ might alter the destructive course of RA.

ELIGIBILITY:
Inclusion Criteria:

(i) Signed informed consent in accordance with applicable regulations

(ii) Males and females aged 21 to 70 years inclusive

(iii) Must have failed at least one DMARD

(iv) Rheumatoid Arthritis fulfilling 1987 ACR revised criteria

(v) Active RA as defined by:

* ≥6 swollen and ≥9 tender joints
* CRP ≥0.8 mg/dL or morning stiffness ≥45 minutes

(vi) If female and of child bearing potential, she must:

* have a negative serum pregnancy test, and
* be using two forms of an effective method of contraception (one form being a barrier method) or be surgically incapable of bearing children or abstinent.

If male and heterosexual, he must:

* agree to use condoms with spermicide throughout the study and for at least 12 weeks following the last infusion.
* vasectomy is an acceptable form of contraception for males and partners of females

(vii) Adequate venous access as defined by the Principal Investigator

(viii) If taking non-steroidal anti-inflammatory medications, must be on stable regimen for four weeks prior to the Screening visit

(ix) If taking prednisone (≤ 10 mg) or equivalent, must be on stable regimen for four weeks prior to Screening visit

Exclusion Criteria:

(i) Prior or current treatment with alkylating agents, or radiation

(ii) Treatment with colchicine within six months prior to Screening

(iii) Experimental anti-rheumatic drugs within 90 days (or five half-lives, whichever is longer) prior to screening

(iv) DMARD therapy four weeks prior to Baseline visit

(v) Intra-articular corticosteroids four weeks prior to the Screening visit

(vi) Bedridden or wheelchair bound patients

(vii) Pregnant or lactating females

(viii) Interstitial lung disease

(ix) Clinically significant cardiac risk factors, including a history of congestive heart failure, angina, and myocardial infarction within the previous six months

(x) History of malignancy, except (a) basal cell carcinoma of the skin and in situ cervical carcinoma that have been excised with no recurrence or treatment within the last five years, and (b) low-grade prostate cancer

(xi) Major organ allograft, or uncontrolled cardiac, hepatic, pulmonary, renal or central nervous system disease, know clotting deficiency, or any illness that increases undue risk to patient

(xii) History of anaphylactic reactions

(xiii) WBC count <4,000/mm3; Neutrophils <2,000/mm3; Platelet count <125,000/mm3; hemoglobin <9g/dL; creatinine >1.4 times the upper limit of normal; liver function test >1.2 times the upper limit of normal

(xiv) Presence of Hepatitis B Surface antigen (HbsAg), Hepatitis C antibody (HCVAb), and/or Hepatitis C quantitative assay, or history of hepatitis (such as autoimmune hepatitis) within one year prior to Screening

(xv) Presence of any confounding illness or syndromes that may interfere with proper evaluation of efficacy, such as other autoimmune disease, psoriatic arthritis, lupus or scleroderma

(xvi) Patients determined by the investigator (e.g., because of known or probable alcohol or drug abuse) to be unreliable for follow-up

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-09; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Denver Arthritis Clinic, Denver, Colorado
  - Radiant Research, Daytona Beach, Florida
  - Ocala Rheumatology Research Center, Ocala, Florida
  - Tampa Medical Group Research, Tampa, Florida
  - Indiana University, Indianapolis, Indiana
  - Arthritis & Rheumatology Clinic of Kansas, Wichita, Kansas
  - Arthritis Center of Reno, Reno, Nevada
  - Altoona Center for Research, Duncansville, Pennsylvania

REFERENCES:
- See also: Click here for more information about this study: A Phase 2, Open-Label, Clinical Study Using Intravenous Paxceed to Treat Patients with Rheumatoid Arthritis — http://www.angiotec.com/clinical/clinical_studies.php